CLINICAL TRIAL: NCT06700525
Title: StandUPTV Habits: Feasibility Trial for Maintaining Reductions in Sedentary Screen Time
Acronym: SUTV Habits
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: California Polytechnic State University-San Luis Obispo (Other); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Chad Stecher@asu.edu, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00020613; 1R01DK135488-01A1 (NIH)
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Sedentary Behaviors; Screen Time; Physical Activity; Glucose Metabolism; Sleep Quality; HbA1c Level
Keywords: sedentary behavior; action planning; evening sedentary screen time; mHealth
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will not have access to study arm assignment and participants will be encouraged not to divulge their study arm assignment during assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- StandUPTV only (Experimental): The StandUPTV application is used to monitor and reduce sedentary screen time (SST). The StandUPTV app has three components: LOCKOUT: Electronic lockout turns off screens when a predetermined limit is reached (50% of baseline value of weekly sedentary screen time). The app also includes planning tools and personalized strategies to limit SST. TEXT: Push notification prompts provide reminders, coaching, and personalized feedback (up to 2 per day). EARN: Opportunities to earn SST by engaging in MVPA, measured in 10-minute bouts.
  Interventions: Behavioral: Non-Sedentary Behavior Habit Formation
- StandUPTV + Action Plans (Experimental): Combining the StandUPTV application with personalized action plans to enhance the maintenance of reduced eSST. At baseline, participants will receive Action Planning Education, action planning worksheet, and weekly personalized text messages reinforcing the action plan. Participant will then receive a daily StandUPTV alert after performing 30 minutes of eSST, and they have 60 minutes after the alert to engage in their active chosen non-sedentary behavior. Financial Incentives: Participants can earn up to $30 per month during the 4-month intervention by starting 10 minutes of their non-sedentary replacement behavior within 60 minutes of the alert. Participants start with $30 in their account and lose $2 for each day they do not perform the behavior. Notifications will be sent via SMS and the StandUPTV app.
  Interventions: Behavioral: Non-Sedentary Behavior Habit Formation; Behavioral: Sedentary Screen Time Reduction Smartphone App

INTERVENTIONS:
Behavioral: Non-Sedentary Behavior Habit Formation — Action Plans Addition to the StandUPTV platform:
  The StandUPTV mHealth platform will be used to assess SST and deliver behavior change components. Participants will receive a technology kit including a Fitbit Charge 4+ and Wi-Fi-enabled smart plugs. The Fitbit and smart plugs will need to be used for the entire duration of the study participation. Participants will also be assisted with establishing an action plan for a non-sedentary break from evening sedentary screen time, which will be trigger by a StandUPTV alert delivered after performing 30 minutes of evening sedentary screen time.
Behavioral: Sedentary Screen Time Reduction Smartphone App — The StandUPTV application is used to monitor and reduce sedentary screen time (SST). The StandUPTV app has three components: LOCKOUT: Electronic lockout turns off screens when a predetermined limit is reached (50% of baseline value of weekly sedentary screen time). The app also includes planning tools and personalized strategies to limit SST. TEXT: Push notification prompts provide reminders, coaching, and personalized feedback (up to 2 per day). EARN: Opportunities to earn SST by engaging in MVPA, measured in 10-minute bouts.
  Arms: StandUPTV + Action Plans

SUMMARY:
Our goal in this study is to further refine StandUPTV, an application designed to reduce SST in adults in our first study (ASU IRB # STUDY00012109), for the StandUPTV Habits program. This program aims to establish a non-sedentary habit triggered by an alert from the StandUPTV application after participants engage in approximately 30 minutes of SST in the evening.

DETAILED DESCRIPTION:
This mobile health (mHealth) pilot study aims to develop and test an intervention designed to maintain reductions in evening sedentary screen time (eSST) over a 12-month period. The study will target a nationally recruited sample of adults at risk for type 2 diabetes and will employ a novel habit formation strategy to address individual barriers to sustained behavior change. As a Phase II pilot study within the ORBIT Model framework, this research seeks to provide critical insights into the relationship between maintained reductions in eSST and metabolic health. The intervention combines theory- and evidence-based approaches, leveraging commercially available screen time monitoring tools to scale the StandUPTV application. This pilot study will lay the groundwork for a subsequent Phase III fully-powered randomized clinical trial, aiming to evaluate the impact of sustained eSST reduction on diabetes and cardiovascular disease risk in a national sample.

ELIGIBILITY:
Inclusion Criteria:

* Insufficiently active as defined by not meeting current US National Guidelines for Physical Activity of 150 minutes of MVPA/week (Measured by the Stanford
* Leisure-Time Activity Categorical Item)
* > 3 hours of SST per day
* Use Android (8.0+) smartphone (8.0+ represents 95% of Android device coverage per https://apilevels.com/)
* Have regular broadband internet in their home or an unlimited data plan
* Able to read/understand English (>5th grade literacy)
* Willing to download StandUPTV Habits
* Willing to wear activPAL and CGM device during study assessment periods
* Willing to have data shared in de-identified form in Dexcom Clarity platform
* Willing to be randomized to either study condition
* Not traveling overnight or longer in the next 4 months

Exclusion Criteria:

* Planned relocation
* Current smoker
* Have a major illness (e.g., heart disease, cancer, renal disease) for which MVPA is contraindicated
* Diagnosed with diabetes or gestational diabetes in the past
* Currently using a CGM
* Pregnant
* Occupation that requires substantial use of personal device for media-related activities (e.g., social media)
* Drug abuse
* Serious psychological disorder
* Not willing to use Fitbit or smart plugs for calculation of sedentary screen time for functionality of StandUPTV app

Ages: 23 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Changes in Sedentary Screen Time | Baseline, 4 months, 12 months
  Minutes per week as measured by Stand UPTV app and activPAL

SECONDARY OUTCOMES:
Changes in moderate to vigorous physical activity | Baseline, 4 months, 12 months
  Minutes per week as measured by activPAL
Changes in Sleep Quality | Baseline, 4 months, 12 months
  Measured in minutes of deep sleep
Changes in Glucose Metabolism | Baseline, 4 months, 12 months
  Measured HbA1c levels
HbA1c Level | Baseline, 4 months, 12 months
  Participants continuous glucose monitoring data will be used to estimates HbA1c levels

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arizona State University, Tempe, Arizona
  - California Polytechnic University San Luis Obispo, San Luis Obispo, California

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share de-identified data on participants sedentary screen time and intervention arm, along with some demographic information and all other outcomes assessed, such as glucose metabolism and sleep.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The investigators will share de-identified data as soon as possible, and no later than the end of the study period. Study data deposited in the ASU Research Data Repository and code deposited in GitHub will be available to the research community in perpetuity.
Access Criteria: Anyone will have access to the de-identified data from this study. The investigators will identify where the data will be available and how to access the data in any publications and presentations that the investigators author or co-author about these data, as well as acknowledge the repositories and funding source in any publications and presentations. The ASU Research Data Repository provides a permanent digital identifier for research data, which complies with NIH data sharing policies. Our analytic code on GitHub can be found by searching for "StandUPTVHabits" on GitHub.
URL: https://dataverse.asu.edu/